CLINICAL TRIAL: NCT01099800
Title: Asthma Disparities in Latino Children:Acculturation,Illness Representations & CAM
Status: Completed | Type: Observational
Sponsor: Arizona State University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); Phoenix Children's Hospital (Other); Scottsdale Healthcare (Other); Albert Einstein College of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 1R01AT005216-01 (NIH); 1R01AT005216-01 (NIH)
Record Dates: First submitted 2010-04-06; First posted 2010-04-08 (Estimated); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Asthma
Keywords: asthma; health disparities; illness representations; CAM; Latino
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Mexican/Mexican American families: Parents and children who self-identify as being of Mexican heritage whether US-born or Mexican-born
- Puerto Rican families: Parents and children who self-identify as Puerto Rican whether US-born or island-born.

SUMMARY:
This interdisciplinary multi-level study moves the research in asthma health disparities from descriptive studies of individual constructs and contexts to testing an integrated, multi-factorial model among Latino families and children with asthma. The investigators seek to gain a more thorough understanding of the interaction of individual characteristics, cultural and experiential factors, social-environmental context, and healthcare system factors on parents' illness representations, use of CAM and controller medications, and children's asthma health outcomes.

This will be a one-year longitudinal, multi-site (Phoenix, AZ and Bronx, NY) study among samples of Mexican (N=300) and Puerto Rican (N=300) parents and children aged 5-12 who have asthma.

Aim #1: Are there differences in illness representations between Mexican and Puerto Rican parents due to social and contextual factors (i.e., acculturation, education, parental age, poverty, child's illness duration, household members with asthma, and parent-healthcare provider relationship)?

Aim #2: Are disparities in asthma control between Mexican and Puerto Rican children due to differences in parents' treatment decisions (CAM and controller medication use) and changes in illness representations over a one year period after controlling for the effects of acculturation, social and contextual factors, environmental triggers, and advice received from others?

DETAILED DESCRIPTION:
Racial and ethnic disparities in asthma health outcomes have been increasing in the United States. These disparities are so striking that researchers and public health officials have issued a call for action to understand why this is occurring. Compared with non-minority children, minority children use controller medication less often, have less continuity of care, and visit emergency departments more frequently. Especially noteworthy has been the increasing prevalence of asthma among Latino (primarily Puerto Rican) children. Individuals of Mexican and Puerto Rican origin constitute 73% of the Latino population in the U.S. and although these two groups share similar historical origins and cultural values, significant heterogeneity exists. Researchers have tended to study Latinos as a single group but recent descriptive asthma research has confirmed differences among Latino subgroups related to prevalence, mortality and morbidity, illness beliefs, and asthma healthcare practices. Puerto Rican children exhibit the highest rates of asthma prevalence and mortality among all ethnic groups while Mexican children have the lowest rates. Asthma disproportionately affects Puerto Rican children: the adjusted odds ratio for lifetime diagnosis compared to non-Latino white children is 2.33. Genetic, environmental, healthcare system and provider factors cannot totally explain the difference in outcomes between these two groups.

Not well examined is the role that culture, acculturation, and illness representations (the way the parent interprets health and illness which influences how he/she manages the child's asthma) may play in parents' asthma treatment decisions and ultimately, children's asthma control. Parental illness representations may account for the differences in the use of complementary and alternative medicine (CAM), inhaled or oral corticosteroids, and leukotriene antagonists that have been observed between Puerto Rican and Mexican families. Acculturation may also play a role in asthma health outcomes. Less-acculturated Mexican families, even if they have known risk factors for poor health outcomes, have better outcomes than more acculturated families. Emerging evidence suggests that acculturation has opposite effects for Puerto Rican versus Mexican children with asthma. U.S. birthplace and higher acculturation among Mexican children is associated with greater risk for asthma and wheezing, while higher acculturation may be protective for Puerto Rican children in terms of diagnosis of asthma and medication adherence.

The past three decades have seen a shift in approaches to studying health and illness behavior from disease-oriented medical models to integrated bio-psycho-social models. The factors leading to asthma health disparities between Mexican and Puerto Rican children are complex and not well understood. Illness representations, the associated treatment decisions (CAM and controller medication use), and the influence of acculturation on these processes, are three factors requiring additional scrutiny. The Common Sense Model of Illness Representation is an integrated model that takes into account environmental, social, and cultural factors as well as patients' beliefs about health and illness. Because parents are the gatekeepers for their children's healthcare and ultimately make the final treatment decisions, it is parents' representation of their children's illness that influences treatment decisions and children's asthma health outcomes.

Before developing interventions that target asthma health disparities among this diverse group of Latino families, it is necessary to gain a more thorough understanding of the interaction of individual characteristics, cultural and experiential factors, social-environmental context, and healthcare system factors. The investigators also need to examine how the interaction of these factors impacts parents' illness representations, use of CAM and controller medications, and children's asthma health outcomes. This innovative study moves the research from descriptive studies of individual constructs and contexts to testing an integrated, multi-factorial model. Targeted interventions, aimed at reshaping illness representations, can be developed and implemented to integrate the family's ethnomedical belief system (medical system based on the cultural beliefs of specific ethnic groups) into the biomedical model. The proposed interdisciplinary multi-level study will address gaps in the evidence base and expand the framework for assessing disparities in asthma health outcomes among Latino children. This will be a one-year longitudinal, multi-site study among samples of Mexican and Puerto Rican parents and children aged 5-12 who have asthma. This age range was selected because children in this age group typically have not assumed daily control for managing their asthma.

The findings from this study will contribute to the knowledge base on the similarities and differences that exist between Mexican and Puerto Rican families regarding asthma illness beliefs and management strategies, and how acculturation influences these factors. Healthcare providers, regardless of their practice setting, can best treat children with asthma if they understand what beliefs parents hold about what causes asthma, the nature of asthma symptoms, its course of action (chronic versus episodic), medications and alternative therapies used in treatment, and expectations for symptom resolution. If parents' beliefs are discordant with the HCPs' beliefs and are not addressed when devising the management plan, there is increased risk for nonadherence. Healthcare providers would also do well to educate themselves as to what CAM therapies parents are using to treat their children's asthma. By doing so, they can then take the lead in eliciting information on CAM use during their contacts with parents to ensure safety when these therapies are used, to educate parents about the advantages and disadvantages of individual CAM therapies, to provide culturally competent care, and to improve adherence to the prescribed medication regimen. If parents feel that they are part of the decision-making process regarding treatment of their children's asthma, they may be more likely to adhere to the prescribed medication regimen. Healthcare providers have an opportunity to intervene at the individual level to effect changes aimed at improving adherence to the prescribed treatment regimen through improved communication, education (both parents and themselves), and partnership with the families.

THEORETICAL FRAMEWORK: A presentation of the theoretical underpinnings and conceptual model for the study is presented here to provide a framework for the discussion of the literature review. The Common Sense Model (CSM) of Illness Representation provides the theoretical framework for investigating the disparities in asthma control through the pathways of parental IR and the use of CAM and controller medications. The model describes a cognitive processing system that includes situational stimuli (perception of the child's symptoms), objective representation of the health threat (illness representation) with its treatment decisions (CAM and controller medication use) and appraisal of the outcomes (asthma control) for the success or failure of those treatment decisions. The model contains a feedback loop with IRs potentially changing over time as the parent gains experience with managing their child's asthma. The three tenets of this model are that the parent is an active problem solver; the IR is the central cognitive construct that drives the parents' treatment decision and appraisal of the outcomes; and IRs are individualized and may not be in agreement with medical facts. The processes of IR, treatment decision, and appraisal of outcomes are shaped by the parent's prior history managing their child's asthma, personality traits, and social and cultural contexts. The social and cultural contexts in which an individual lives play an important role in illness representations in two ways:"1) culture provides the labels for categorizing the events/symptoms that define illness and ensures culturally common views of a given disease or illness; and 2) culture provides social and personal contacts that the parent then uses in constructing the IR and also in developing the action plan for coping with the disease threat." Prior experience with their child's asthma management generates stored memories about the success or failure of the chosen treatment strategy, which can influence how the parent perceives the child's symptoms for the current episode and that treatment decision. There are five distinct attributes of illness representations:

1. identity - the disease label and the somatic symptoms the parent associates with the disease.
2. cause - the parent's ideas about what causes the disease.
3. consequences - the parent's perceived short and long term effects of the disease, and the physical, social, emotional, and economic consequences of the disease.
4. time-line - the parent's expectations about disease duration: acute, chronic, or episodic/cyclical.
5. controllability - the parent's ideas about cure or recovery either through their own actions or medical intervention.

DESIGN: This will be a longitudinal study of parental illness representations and CAM and controller medication use among a diverse sample of 300 Latino families (primarily Mexican and Puerto Rican) of children with asthma aged 5-12. This age range was selected because children in this age group typically have not assumed daily control for managing their asthma. We will use a structured interview with parents, conduct a short interview with the children, obtain objective measures of lung function from the children, and review children's medical records. Interviews and child assessments will be conducted at five time periods: enrollment, and 3, 6, 9 and 12 months after enrollment, for a total data collection period of 12 months. This assessment schedule will allow us to capture seasonal variations in the children's asthma symptoms as well as conform to the recommendation by NAEPP that children on daily controller medications have follow-up visits every 3 months. Medical record abstractions will take place at the 12-month follow-up.

Figure 1. Conceptual framework and proposed relationships

Sample and Setting: To ensure diverse representation of Latino families and healthcare settings, the sample will be recruited from two school-based health clinics and one clinical practice site in Phoenix, AZ, and two inner-city hospital asthma clinics in the Bronx, NY. A multisite study is warranted because neither site alone has sufficient numbers of both Mexican and Puerto Rican families to conduct this research independently. It is also preferable that interviews and assessments be conducted simultaneously among these two populations to minimize seasonal variations in asthma symptom severity and control and to maximize standardization of survey administration across time and samples. Approximately 300 families will be recruited and enrolled from the asthma/allergy and general pediatric clinics and ER at Jacobi Medical Center and North Central Bronx Hospital (N= 150), Phoenix Children's Hospital Breathmobile (N= 75), and the two school-based health clinics in Phoenix (N= 75). These clinical partner sites provide adequate populations of inner-city, poor Mexican and Puerto Rican children with asthma to recruit the study sample, thus we anticipate no problems recruiting and enrolling 300 families.

Prescreening: Approximately 400 parents and children with asthma aged 5-12 years old will be invited to participate in the study if they meet the eligibility criteria below. Our previous research studies yielded refusal rates ranging from 15% to 30%. We have assumed a conservative 20% refusal rate, which will yield approximately 300 families agreeing to participate in the study.

Eligibility criteria: a) The child must be between 5 and 12 years of age, b) have a diagnosis of asthma (described below) as obtained from the child's medical record, c) the family is Latino (English or Spanish speaking) as self-identified by the primary caregiver, d) the child has no other significant pulmonary conditions (e.g., cystic fibrosis), e) the participating parent has primary or at least equal responsibility for the day-to-day management of the child's asthma, and f) no cognitive learning disability that could interfere with the parent's or child's (as determined by parents' report) ability to comprehend the interview questions. All of the recruitment sites have computerized data systems that allow participant identification by diagnosis, age, and ethnicity. If no documentation of a diagnosis of asthma is found in the medical record but asthma is suspected, the potential participant will be offered an appointment for a bronchodilator test for the child. Prior to the test date, the potential participants will be instructed to withhold short-acting β2- agonist medications (e.g., albuterol), caffeine, medicines and drinks containing methylxanthines (e.g., root beer), long-acting bronchodilator medications (e.g., salmeterol, formoterol), and combination agents (e.g., Advair, Symbicort) for 24 hours. Herbal preparations (e.g., kanpo, ding chan tang) and over-the-counter medications (e.g., Primatene™ mist) affecting pulmonary function will also be restricted accordingly.

Multiple Children in One Family: It will be explained to the primary caregiver that only one child may participate in this study. If more than one child meets the criteria and is interested, the RA will put the names of those children who are interested into a hat and randomly pull one name out of the hat to identify who will be the subject.

INFORMED CONSENT: The goal will be to enroll the parent who assumes primary or at least equal responsibility for the day-to-day management of the child's asthma. Written consent will be obtained by the RNA from the parent for (a) conducting the parental interview, (b) abstracting pre-identified data from the child's medical record data, and (c) obtaining permission to interview the child and have the child perform the spirometry maneuver. Verbal assent from the child to complete the interview and spirometry maneuver will also be obtained by the RNA. Subjects will be informed that they are free to withdraw from the study at anytime, that nonparticipation will not affect their or their children's healthcare, and that their names will not appear on study materials. We will use a unique 4-digit number to code their data and provide confidentiality. All consent and assent materials will be available in English and Spanish. Parents will decide which language they prefer.

STATISTICAL MODELS AND METHODS OF ANALYSIS: Eligible participants who decline to participate will be compared with those enrolled on demographic characteristics to check for sample bias. Descriptive statistics will be used to identify the distribution of data and total instrument scale scores for each of the study surveys. Means and standard deviations will be examined for continuous variables and proportions for categorical variables. Linear regression (SAS) will be used to examine Aim 1 of the study. A growth model with time varying covariates (using MPlus) will be used to examine Aim 2 of this study. Growth modeling allows for examination of individuals over time on one or more outcome variables (e.g., IRs, treatment decisions, and asthma control). Random effects are specified in the model to capture individual differences in development. MPlus uses a multivariate approach and maximum likelihood estimation for this type of model. The time scores for the slope growth factor are fixed to 0, 1, 2, 3, and 4 to define a linear growth model with equidistant time points. The zero time score for the slope growth factor defines the intercept growth factor, the coefficients of the intercept growth factor are fixed at one, the residual variances of the outcomes are estimated and allowed to be different across time, and the residuals are not correlated. Illness representations, CAM, and controller medication use are time varying variables in the model.

Data reduction: Psychometric analyses will be conducted for the AIRS©, C-ACT, P-CASCL/CASCL scales separately for each ethnic group to determine if the factor structure (construct validity), internal consistency (reliability), and external validity is replicated from the original instrument across these Latino subgroups. Internal consistency for all scales will be assessed using Cronbach's alpha. Factor analyses will be conducted specifying varimax rotation and a minimum eigenvalue of 1. External validity for the AIRS© instrument will be assessed by testing the hypotheses from the original development work which showed that scores on the AIRS© instrument differed by ethnicity, education, and poverty and that it differentiated children on an appropriate versus suboptimal medication regimen.

Missing Data: We recognize the drawback of only analyzing cases with complete data. Our primary strategy will be to minimize attrition to the greatest extent possible. Growth models allow for missing data on the dependent variable using full maximum likelihood (FIML) methods which assume that the data are missing at random and that dependent variable scores tend to be correlated with the previous measure from earlier data collection points. When predictor variables are missing, the investigators will use multiple imputation. For the multiple imputations, the investigators will utilize a Markov Chain Monte Carlo method to impute enough data to have a monotone missing data pattern. Once the investigators have a monotone missing data pattern, the investigators will employ imputation approaches appropriate for the type of data (continuous, dichotomous, or low frequency count data). We will perform sensitivity analyses to ensure that results are similar under various assumptions. Ultimately, the investigators will determine whether imputation is valid and has sufficient added value with our data to justify the complexity involved in reporting these analyses.

Non-normal Distributions: Full attention will be given to the distributional properties of variables and to regression diagnostics. We will employ negative binomial error assumptions and make adjustments for outlying data points.

STATISTICAL ANALYSIS Aim #1: Are there differences in illness representations between Mexican and Puerto Rican parents due to social and contextual factors (i.e., acculturation, education, parental age, poverty, child's illness duration, household members with asthma, and parent-healthcare provider relationship)? Ethnicity (0=Mexican 1=Puerto Rican) and healthcare setting (1=school-based 2=Breathmobile 3=hospital-based) will be entered as classification factors in the regression model with the above covariates to examine differences in the total AIRS© score as well as the individual subscale scores. The interaction of acculturation and ethnic group will be included to assess the potential mediation effect of acculturation on IR.

Aim #2: Are disparities in asthma control between Mexican and Puerto Rican children due to differences in parents' treatment decisions (CAM and controller medication use) and changes in illness representations over a one year period after controlling for the effects of acculturation, social and contextual factors, environmental triggers, and advice received from others?

There will be a maximum of 5 observations on each subject in the sample (over the 5 time periods). The primary interest is in the regressions of asthma control on time of assessment. The model includes these regressions with the parameters assumed to be fixed; these fixed regressions will be specified separately by ethnic group. The test of homogeneity of these regressions will be a primary research interest. Non-homogeneity of these regressions would suggest ethnic group differences in the relationship between time and asthma control. Individual regressions of asthma control on time for each subject will also be included in the model. These regressions will be random because they are associated with levels of a random factor (subjects). They can be regarded as deviations from the overall fixed regression. Henderson202 discusses methods for random regressions and the assumptions regarding them; the analysis of mixed models (fixed and random effects) of this type, and tests of homogeneity of regressions in mixed models. Because the investigators hypothesize that the level of acculturation could potentially influence the results, it will be included as a covariate in the model. Following conventions outlined by Kline,Byrne,and Cudeck & Browne,our criteria for assessing adequacy of fit will be: chi-square to df ratio of less than 2, comparative fit index (CFI) and Tucker-Lewis Index (TLI) at or above .90, and a root mean square error approximation (RMSEA) at or below .08.

Examination of Mediation. We will examine mediation in models with structural equations, testing the significance of direct and indirect effects and their equality. Testing will be by the delta method or bootstrapping. While tests involving indirect effects are of primary interest, the investigators will in some cases carry out a priori tests reflecting Mackinnon's recommendations. Mediation will be tested through first showing that X (e.g., ethnic group) is associated with both M (e.g., illness representation) and Y (e.g., treatment decision). Second, a path model is estimated by simultaneously regressing (a) Y on M and X, and (b) M on X. This will be repeated specifying X=illness representation, M=treatment decision, and Y=asthma control. The paths from X to M and from M to Y must each be statistically significant by this criterion, in addition to the significance of the indirect effect. If the path from X to Y drops to zero, full mediation is suggested. Partial mediation is suggested to the extent that X still predicts Y with the mediator(s) simultaneously entered. These first-stage tests also result from the model estimation used for testing the indirect effect. In that model estimation, the investigators use full information methods (e.g., FIML) unless there is clear indication that OLS is adequate. Henderson and Ceci describe delta-test methods for moderation and mediation.

ELIGIBILITY:
Inclusion Criteria:

* child must be between 5 and 12 years of age,
* have a diagnosis of asthma as obtained from the child's medical record,
* the family is Latino (English or Spanish speaking) as self-identified by the primary caregiver,
* the child has no other significant pulmonary conditions (e.g., cystic fibrosis),
* the participating parent has primary or at least equal responsibility for the day-to-day management of the child's asthma, and
* no cognitive learning disability that could interfere with the parent's or child's (as determined by parents' report) ability to comprehend the interview questions.

Exclusion Criteria:

* children not meeting the above inclusion criteria
* parents who do not have primary or equal responsibility for the child's asthma mangement

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: To ensure diverse representation of Latino families and healthcare settings, the sample will be recruited from two school-based health clinics and one clinical practice site in Phoenix, AZ, and two inner-city hospital asthma clinics in the Bronx, NY. Approximately 300 families will be recruited and enrolled from the asthma/allergy and general pediatric clinics and ER at Jacobi Medical Center and North Central Bronx Hospital (N= 150), Phoenix Children's Hospital Breathmobile (N= 75), and the two school-based health clinics in Phoenix (N= 75).
Sampling Method: Non-Probability Sample
Enrollment: 534 (Actual)
Dates: Start 2010-06-23 (Actual); Primary Completion 2014-08-25 (Actual); Study Completion 2014-08-25 (Actual)

PRIMARY OUTCOMES:
asthma control | basline, 3,6,9, and 12 months
  Level of asthma control will be assessed per NAEPP guidelines which incorporate a structured assessment of symptoms and spirometry.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly J Sidora-Arcoleo, PhD, MPH, Principal Investigator — Arizona State University
Locations (4):
- United States (4):
  - Arizona State University College of Nursing and Health Innovation, Phoenix, Arizona
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Scottsdale Healthcare NOAH Clinic, Scottsdale, Arizona
  - Yeshiva University, The Bronx, New York

REFERENCES:
- [Derived] Arcoleo K, Marsiglia F, Serebrisky D, Rodriguez J, Mcgovern C, Feldman J. Explanatory Model for Asthma Disparities in Latino Children: Results from the Latino Childhood Asthma Project. Ann Behav Med. 2020 Mar 24;54(4):223-236. doi: 10.1093/abm/kaz041. PMID 31586174
- [Derived] Arcoleo KJ, McGovern C, Kaur K, Halterman JS, Mammen J, Crean H, Rastogi D, Feldman JM. Longitudinal Patterns of Mexican and Puerto Rican Children's Asthma Controller Medication Adherence and Acute Healthcare Use. Ann Am Thorac Soc. 2019 Jun;16(6):715-723. doi: 10.1513/AnnalsATS.201807-462OC. PMID 30860858